CLINICAL TRIAL: NCT05235711
Title: The Role of Interferon-gamma in Immune Responses to Invasive Candidiasis
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Paschalis Vergidis, Principal Investigator, Mayo Clinic
Other Study IDs: 21-008735
Record Dates: First submitted 2022-01-04; First posted 2022-02-11 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Fungal Infection; Candidiasis
MeSH Terms: conditions — Mycoses; Candidiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum/plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of the study is to investigate the role of the human immune response to candidemia/invasive candidiasis as it relates to the cytokine interferon-gamma.

DETAILED DESCRIPTION:
In this study, patients with Candida bloodstream infection, peritonitis/intra-abdominal abscess, and pleural empyema will be enrolled.

Persistent candidiasis confirmed by culture will be defined as follows: (i) Candida bloodstream infection present for >48 hours after initiation of effective antifungal treatment and after removal of intravenous devices, (ii) Intra-abdominal infection (peritonitis or abscess) that persists for >96 hours after source control intervention and effective antifungal treatment, (iii) Pleural empyema that persists for >96 hours after placement of drainage catheter and effective antifungal treatment.

Outcomes in patients with and without persistent candidiasis will be assessed.

ELIGIBILITY:
Subjects must meet all following inclusion criteria to qualify for the study:

1. Willing and able to provide written informed consent. If the subject is unable to consent for himself/herself, a legally authorized representative must provide informed consent on his/her behalf.
2. Males or females ≥18 years of age
3. Patients having one or more systemic signs attributable to candidemia or invasive candidiasis (fever, hypothermia, hypotension, tachycardia, tachypnea, local signs of inflammation).
4. Isolation of Candida from blood, intra-abdominal abscess/peritoneal fluid or pleural fluid.

Exclusion Criteria

Subjects must NOT meet any of the following exclusion criteria to qualify for the study:

1. Severe neutropenia (absolute neutrophil count <500 cells/microL)
2. Profound lymphopenia (<300 cells/microL)
3. The Principal Investigator (PI) is of the opinion the subject should not participate in the study.
4. Females who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Candida bloodstream infection, peritonitis/intra-abdominal abscess, and pleural empyema
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 30 days
  All-cause mortality

SECONDARY OUTCOMES:
Serum concentration of IFN-gamma and other cytokines by multiplex ELISA | 1 week
  Serum concentration of IFN-gamma and other cytokines by multiplex ELISA
Plasma IFN-gamma concentration after dual innate and adaptive immune system stimulation by QuantiFERON Monitor assay | 1 week
  Plasma IFN-gamma concentration after dual innate and adaptive immune system stimulation by QuantiFERON Monitor assay
Intracellular expression of IFN-gamma expression by a CD8 T-cell competence assay | 1 week
  Intracellular expression of IFN-gamma expression by a CD8 T-cell competence assay
In vitro antifungal activity of polymorphonuclear leukocytes in the presence or absence of interferon-gamma by colorimetric method | 1 week
  In vitro antifungal activity of polymorphonuclear leukocytes in the presence or absence of interferon-gamma by colorimetric method

CONTACTS AND LOCATIONS:
Overall Officials: Paschalis Vergidis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinical Trial — https://www.mayo.edu/research/clinical-trials/cls-20526487